CLINICAL TRIAL: NCT06543901
Title: Comparative Study Between (MIPO)Submuscular Plate Fixation of Fracture Femur and Conservative Management With Thomas Splint in Children From 5 to 8 Years Old: A Randomized Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Omar Sabry, Dr., Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-321-2021
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Femur Fracture
MeSH Terms: conditions — Femoral Fractures | interventions — Traction

STUDY DESIGN:
Intervention Model Description: This study employs a parallel-group randomized controlled trial (RCT) design. In this model, participants are randomly assigned to one of two groups: the intervention group or the control group. Each participant remains in their assigned group for the duration of the study, receiving either the intervention being tested (MIPO submuscular plate fixation) or the control treatment (conservative management with Thomas splint). This design allows for a direct comparison of the outcomes between the two groups, minimizing bias and ensuring the reliability of the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Submuscular plate (Experimental): The patient underwent open reduction and internal fixation by being fixed with a submuscular plate
  Interventions: Procedure: Submuscular plating
- traction with a thomas splint and then casting (Active Comparator): the patient was placed on traction with a thomas splint and then was casted in a spica cast
  Interventions: Procedure: Traction and casting

INTERVENTIONS:
Procedure: Submuscular plating — the patient was fixed with a submuscular plate
  Arms: Submuscular plate
Procedure: Traction and casting — the patient was placed on a traction with a thomas splint and then was casted with a hip spica
  Arms: traction with a thomas splint and then casting

SUMMARY:
This randomized clinical study compares the outcomes of two treatment methods for femur fractures in children aged 5 to 8 years: Minimally Invasive Plate Osteosynthesis (MIPO) using submuscular plate fixation and conservative management using a Thomas splint. The study evaluates the efficacy, safety, and recovery outcomes of both techniques. Key parameters include healing time, functional outcomes, complication rates, and patient and caregiver satisfaction. The findings aim to provide evidence-based recommendations for the optimal management of femur fractures in young children, balancing the benefits and risks of surgical versus non-surgical approaches.

DETAILED DESCRIPTION:
Introduction:

Femur fractures are common pediatric injuries that require effective treatment to ensure proper healing and prevent long-term complications. While conservative management with a Thomas splint is a traditional method, Minimally Invasive Plate Osteosynthesis (MIPO) using submuscular plate fixation has gained popularity due to its potential for faster recovery and reduced complications. This study aims to compare the outcomes of these two treatment modalities in children aged 5 to 8 years.

Objectives:

To compare the healing time between MIPO submuscular plate fixation and conservative management with Thomas splint.

To assess the functional outcomes of both treatment methods. To evaluate the complication rates associated with each treatment. To measure patient and caregiver satisfaction with each treatment approach.

Methods:

Study Design: Randomized clinical study. Participants: Children aged 5 to 8 years with femur fractures, meeting specific inclusion and exclusion criteria.

Randomization: Participants will be randomly assigned to either the MIPO submuscular plate fixation group or the conservative management with Thomas splint group.

Interventions:

MIPO Group: Surgical intervention using minimally invasive techniques to place a submuscular plate for fracture fixation.

Thomas Splint Group: Conservative management using a Thomas splint for immobilization and fracture healing.

Follow-Up: Regular follow-up visits at specified intervals to monitor healing, assess functional outcomes, and record any complications.

Outcome Measures:

Primary Outcome: Healing time, defined as the time from intervention to radiographic evidence of fracture union.

Secondary Outcomes:

Functional outcomes assessed using standardized pediatric orthopedic scoring systems.

Complication rates, including infection, malunion, nonunion, and reoperation rates.

Patient and caregiver satisfaction assessed through questionnaires and interviews.

ELIGIBILITY:
Inclusion Criteria:

1. Children from 5 to 8 years.
2. Patients with midshaft or distal shaft femur fracture.
3. Fracture pattern: transverse - oblique - spiral.
4. Children must be < 45 KG.

Exclusion Criteria:

1. Open fracture
2. Any associated fracture in the same limb or in contralateral limb
3. Associated serious internal organ injury or vascular injury
4. Proximal, distal physeal femur fracture.
5. Patient with pathological bone disease as osteogenesis imperfecta.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Bony union | 6 weeks and 12 weeks
  we do sequential xrays until we can see a bony union

SECONDARY OUTCOMES:
Any associated complications | 6 weeks and 12 weeks
  such as pain, infection or failure of reduction

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy Hospital - Faculty of Medicine - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes